CLINICAL TRIAL: NCT06139133
Title: The Impact of Vitamin D Supplementation on Gestational Diabetes Mellitus Risk in Pakistani Females: A Randomized Controlled Trial.
Brief Title: The Impact of Vitamin D Supplementation on Pregnant Women With the Risk of GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IIMC, Riphah International University, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Riphah/IIMC/IRC/23/3073
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Mellitus; Pregnancy; High risk women; Vitamin D supplementation
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo supplementation Group (Placebo Comparator): Pregnant women with 07-11 weeks of gestation having normal response to 75g OGTT but with low levels of Vitamin D3 (<30ng/ml) will be included. The study subjects will be randomly assigned to receive placebo until delivery.
  Interventions: Drug: Placebo supplementation
- Vitamin D supplementation group (Experimental): pregnant women with 07-11 weeks of gestation having normal response to 75g OGTT but with low levels of Vitamin D3 (<30ng/ml) will be included for Vitamin D3 supplementation (2 00,000 IU/Week) for 04 -06 week. The study subjects will be randomly assigned to receive vitamin D3 supplementation (2 00,000 IU/Week) for 04 -06 weeks.
  Interventions: Drug: Vitamin D supplementation

INTERVENTIONS:
Drug: Placebo supplementation — Placebo
  Arms: Placebo supplementation Group
Drug: Vitamin D supplementation — Vitamin D3 supplementation (2 00,000 IU/Week)
  Arms: Vitamin D supplementation group

SUMMARY:
A clinical trial will be conducted in Chemical pathology department in collaboration with Gyne &Obs department of PRH, IIMC over a period of 02 years w.e.f. December 15, 2023. 350 pregnant women with 07-11 weeks of gestation and having a high risk for GDM with low Vitamin D3 levels and normal response to 75g OGTT will be randomly assigned to receive either vitamin D3 supplementation (2 00,000 IU/Week) for 04 -06 weeks or Placebo. These women will be checked for the diagnosis of GDM with 75 g OGTT at 24- 28 weeks of gestation. The outcome of the study will be the incidence of GDM based on the International Association of Diabetes and Pregnancy Study Groups Criteria.

DETAILED DESCRIPTION:
Gestational diabetes mellitus is a common condition among pregnant women with metabolic implications for both the mother and offspring. Studies have suggested a potential role of vitamin D status in GDM risk, but evidence from randomized controlled trials is inadequate and inconclusive. A research has been planned to investigate the effect of vitamin D supplementation on GDM development among high risk pregnant women through a well-designed RCT Pregnant women at a risk to develop GDM with low vitamin D levels (<30 ng/mL) at 07-11 weeks of gestation will be recruited and randomly assigned to receive either vitamin D3 supplementation (2 00,000 IU/Week) for 04 -06 weeks or placebo. Randomization will be achieved using a computer-generated random sequence or a randomization table. The allocation will be done in a 1:1 ratio, with equal numbers of participants assigned to the vitamin D and placebo groups. The primary outcome will be the incidence of GDM based on the International Association of Diabetes and Pregnancy Study Groups Criteria after 75 g OGTT.

This study will contribute to the understanding of the relationship between vitamin D and GDM risk through a well-designed RCT with integrated approaches. The findings may inform clinical practice and public health recommendations for vitamin D supplementation during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with 07-11 weeks of gestation
* 21 - 40 Years age range
* Pregnant women with high risk for GDM
* history of GDM in their previous pregnancy,
* one or more first-degree relative diagnosed with diabetes mellitus,
* overweight-BMI >25 kg/m2 or obese-BMI >30 kg/m2 at their first antenatal visit
* with a history of polycystic ovarian syndrome.
* Pregnant women with 07-11 weeks of gestation having normal response to 75g OGTT
* Low levels of Vitamin D3 (<30ng/ml)

Exclusion Criteria:

* Women already diagnosed with diabetes mellitus
* Any other systemic disease.
* High risk pregnant women diagnosed with diabetes on the basis of 75g OGTT
* High risk pregnant women with normal vitamin D3 levels (>30ng/ml).

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes mellitus with 75g OGTT | 28 weeks
  75g-OGTT is an oral glucose tolerance test done by ingesting 75 g glucose dissolved in water in the morning at 7- 8 am.
  * Patient seated quietly & relaxed for 30 mins before taking the test
  * A zero-time (baseline) blood sample is drawn
  * The patient is then given a 75-g glucose solution to drink within 5 minutes
  * 2nd Sample - 1h after consumption of sugar to measure the blood glucose
  * 3rd Sample- 2h after consumption of sugar to measure blood glucose
  * Both blood samples should be kept in fluoride-containing collection tubes
  Interpretation of Test:
  GDM diagnosed if any one of the following is present after 75g OGTT:
  * FPG: >92 mg/dl
  * 1-hour PG: >180 mg/dl
  * 2-hour PG: >153 mg/dl
    * THE WHO GUIDELINES (2018)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Nadim Akbar Khan, FCPS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No